CLINICAL TRIAL: NCT05221957
Title: Effects of Preoperative Correction of Anemia With Intravenously Iron in Colorectal Cancer Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: REG-056-2020
Record Dates: First submitted 2021-04-14; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Cancer; Anemia; Iron-deficiency
Keywords: Anemia; Iron-deficiency anemia
MeSH Terms: conditions — Colorectal Neoplasms; Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: Propensity score matched cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iron(III)isomaltoside 1000 (Experimental): Anemic patients receiving treatment with iron(III)isomaltoside
  Interventions: Drug: Iron(III)isomaltoside
- Historical comparison (No Intervention): Anemic patients without receiving treatment prior to surgery. Historical comparison.
- Concurrent comparison (No Intervention): Non-anemic patients not receiving treatment with iron(III)isomaltoside prior to surgery

INTERVENTIONS:
Drug: Iron(III)isomaltoside — Individual weight and hemoglobin dependent dosage
  Arms: Iron(III)isomaltoside 1000

SUMMARY:
The aim of the study is to examine the effects of anemia correction with intravenous administered iron on clinical outcomes and the immune response on the tumor in patients with planned colonic- or rectal cancer surgery.

The study will be performed as a retrospective propensity score-matched cohort study with an examination of immune response in tumor and clinical outcomes, between patients with anemia without correction with iron(III)isomaltoside, non-anemic patients, and anemic patients treated with iron(III)isomaltoside prior to surgery. Propensity score matching will ensure identification of controls from a pool of patients treated at the Department of Surgery, Zealand University Hospital. The two control groups will be: an anemic historical control group (group 1), and a non-anemic concurrent control group (group 2). Group 3 will be the treatment group, with patients with anemia and treated with iron(III)isomaltoside.

The study period of cases undergoing i.v. treatment will be 1st of February 2017 to 31st of October 2019 with approximately 70 cases included

ELIGIBILITY:
Inclusion Criteria:

* Undergoing curative intended surgery for colon or rectum cancer
* UICC stage I-III

Exclusion Criteria:

* Neoadjuvant oncological treatment
* Acute / subacute surgery
* Palliative surgery
* Other pathology than adenocarcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Gene expression and lymphocyte infiltration of the tumor | 1 day after surgery
  770 gene expression analysis and CD3/CD8+ lymphocyte infiltration of the primary tumor
Complications | 30 days after surgery
  Postoperative complications after surgery measured by the Clavien-Dindo classification

SECONDARY OUTCOMES:
Length of stay | up to 100 days
  Length of postoperative hospital stay, until discharge or death.
Readmission | Within 30 days after surgery
  Any readmission over 24 hours in length
Time to chemotherapy | up to 100 days
  Tme from surgery to adjuvant oncological treatment for patients with high risk stage II and stage III disease
Perioperative blood transfusions | from outpatient assesment to 30 days after surgery
  Any blood transfusions measured in ml.
Mortality | 30 days, 90 days and one year
  Mortality